CLINICAL TRIAL: NCT01481467
Title: Evaluation of a Multi-faceted Influenza Vaccination Implementation Strategy for Health Care Workers in Hospitals
Brief Title: Evaluation of an Influenza Vaccination Implementation Strategy for Hospital Health Care Workers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Josien Riphagen-Dalhuisen, MD, PhD fellow, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 125030012
Record Dates: First submitted 2011-11-10; First posted 2011-11-29 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-12

CONDITIONS: Influenza
Keywords: influenza vaccination; intervention mapping; hospital care; respiratory infections; vaccination
MeSH Terms: conditions — Influenza, Human; Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Influenza vaccination implementation strategy applied.
  Interventions: Behavioral: Influenza vaccination implementation strategy
- Control (No Intervention): Usual care.

INTERVENTIONS:
Behavioral: Influenza vaccination implementation strategy — A multi-faceted influenza vaccination implementation strategy
  Arms: Intervention

SUMMARY:
Influenza is a serious disease which can cause severe illness and even death among patients. Health care workers (HCWs) often get infected with influenza and up to 76% of them keep working while being ill. Immunizing HCWs is therefore an essential factor in protecting patients from influenza as HCWs easily transmit influenza to their patients.

However, despite recommendations from the Dutch Health Council since 2007, vaccine uptake among HCWs remains low.

The aim of this study is to develop an effective implementation strategy on the basis of previous behavioural studies and to evaluate its value in a clustered randomized trial in all Dutch University Medical Centers (UMCs). Also, we want to assess the program elements that are associated with a higher vaccine uptake and the cost-effectiveness of such an implementation strategy.

The results of this study will give more insights in the way influenza vaccination campaigns should be directed in order to achieve high vaccine uptake rates among HCWs in hospitals.

DETAILED DESCRIPTION:
Since influenza vaccination rates among hospital HCWs are low, we developed an implementation program which will be tested in this large target group. The primary objective is to evaluate the short- and long-term effects of a multi-faceted implementation program to improve influenza vaccine uptake among HCWs in hospitals over two influenza seasons. Its clinical effects are assessed by means of a randomized controlled trial in selected divisions (e.g. internal medicine, pediatric ward) of all six randomized UMCs in the Netherlands. Secondary aims are to assess program elements associated with higher vaccine uptake among the target group and to evaluate the cost-effectiveness of the program.

The program will be developed using the Intervention Mapping method taking into account all evidence from systematic literature review and the questionnaire study among HCWs in UMCs as part of our before measurement (2008). The Intervention Mapping method is a theoretical framework developed in the field of health education and promotion to systematically design theory and evidence based health promotion programs.

In 2008, we have selected five divisions of all UMCs that will take part in the trial. Before measurement showed wide variation of uptake (<15-50%) and 11 determinants that explained more than 95% of the vaccination behaviour. Three UMCs will adopt the intervention developed by the research group using the Intervention Mapping method, and three UMCs will serve as controls. The current implemented programs in the UMCs vary widely ranging from passive information systems to involvement of the Board of Directors. Our intervention will exist of a multi-faceted program aimed at both HCWs and management of the divisions. Our primary outcome will be the recorded vaccine uptake among HCWs in the UMCs.

To evaluate the short-term and long-term process of the program, web-based questionnaires will be developed and directed at all health care workers of the selected divisions in all UMCs. The questionnaire will contain questions about vaccine uptake and HCWs' opinions on influenza, vaccination and the vaccination campaign. Absenteeism will also be registered.

Finally, patient data will be collected in the participating divisions of all UMCs in order to investigate if there is a relationship between vaccinating HCWs and morbidity and mortality in patients because of influenza.

ELIGIBILITY:
Inclusion Criteria for clusters:

* University Medical Hospital in the Netherlands

Exclusion Criteria for clusters:

* Absence of consent to be randomized

Inclusion Criteria for participants:

* Health care staff at University Medical Hospitals
* Patients cared for during the study influenza epidemics of selected divisions

Exclusion Criteria for participants:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-12 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Influenza vaccine uptake among health care workers in the UMCs | Up to 2 months
  Influenza vaccine uptake among health care workers of all UMCs. Measured by means of data provided by the departments of occupational health. For the assessment of short-term effects vaccine uptake is measured after the first influenza season (2009/2010) in February-March 2010 and for the long-term effects it is measured after the second influenza season (2010/2011) in March-April 2011.

SECONDARY OUTCOMES:
Absenteeism among health care workers during influenza epidemics | Up to 5 months
  Absenteeism among HCWs is assessed by means of data provided by the department of occupational health at the end of both influenza seasons.
Patient morbidity and mortality | Up to 5 months
  After the second influenza season (2010/2011) patient data are collected from selected departments of both the intervention and control UMCs. It is measured by assessing if patients had influenza, if they were tested on influenza, if they had developed a pneumonia, if they were admissioned to the intensive care unit, the duration of hospitalization and intensive care admission and finally mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Josien Riphagen-Dalhuisen, MD, Principal Investigator — University Medical Centre Groningen/ University of Groningen; Eelko Hak, PhD, Study Director — University Medical Centre Groninge/University of Groningen
Locations (2):
- Netherlands (2):
  - University Medical Centre Groningen, Groningen
  - University Medical Centre, Groningen

REFERENCES:
- [Background] Osterholm MT, Kelley NS, Sommer A, Belongia EA. Efficacy and effectiveness of influenza vaccines: a systematic review and meta-analysis. Lancet Infect Dis. 2012 Jan;12(1):36-44. doi: 10.1016/S1473-3099(11)70295-X. Epub 2011 Oct 25. PMID 22032844
- [Background] Hayward AC, Watson J. Effectiveness of influenza vaccination of staff on morbidity, and mortality of residents of long term care facilities for the elderly. Vaccine. 2011 Mar 16;29(13):2357-8. doi: 10.1016/j.vaccine.2011.01.020. Epub 2011 Feb 2. No abstract available. PMID 21295099
- [Background] Potter J, Stott DJ, Roberts MA, Elder AG, O'Donnell B, Knight PV, Carman WF. Influenza vaccination of health care workers in long-term-care hospitals reduces the mortality of elderly patients. J Infect Dis. 1997 Jan;175(1):1-6. doi: 10.1093/infdis/175.1.1. PMID 8985189
- [Background] Wilde JA, McMillan JA, Serwint J, Butta J, O'Riordan MA, Steinhoff MC. Effectiveness of influenza vaccine in health care professionals: a randomized trial. JAMA. 1999 Mar 10;281(10):908-13. doi: 10.1001/jama.281.10.908. PMID 10078487
- [Background] Carman WF, Elder AG, Wallace LA, McAulay K, Walker A, Murray GD, Stott DJ. Effects of influenza vaccination of health-care workers on mortality of elderly people in long-term care: a randomised controlled trial. Lancet. 2000 Jan 8;355(9198):93-7. doi: 10.1016/S0140-6736(99)05190-9. PMID 10675165
- [Background] Saxen H, Virtanen M. Randomized, placebo-controlled double blind study on the efficacy of influenza immunization on absenteeism of health care workers. Pediatr Infect Dis J. 1999 Sep;18(9):779-83. doi: 10.1097/00006454-199909000-00007. PMID 10493337
- [Background] Weingarten S, Riedinger M, Bolton LB, Miles P, Ault M. Barriers to influenza vaccine acceptance. A survey of physicians and nurses. Am J Infect Control. 1989 Aug;17(4):202-7. doi: 10.1016/0196-6553(89)90129-6. PMID 2774292
- [Background] Christini AB, Shutt KA, Byers KE. Influenza vaccination rates and motivators among healthcare worker groups. Infect Control Hosp Epidemiol. 2007 Feb;28(2):171-7. doi: 10.1086/511796. Epub 2007 Jan 17. PMID 17265398
- [Background] Doebbeling BN, Edmond MB, Davis CS, Woodin JR, Zeitler RR. Influenza vaccination of health care workers: evaluation of factors that are important in acceptance. Prev Med. 1997 Jan-Feb;26(1):68-77. doi: 10.1006/pmed.1996.9991. PMID 9010900
- [Background] Smedley J, Palmer C, Baird J, Barker M. A survey of the delivery and uptake of influenza vaccine among health care workers. Occup Med (Lond). 2002 Aug;52(5):271-6. doi: 10.1093/occmed/52.5.271. PMID 12181376
- [Background] Canning HS, Phillips J, Allsup S. Health care worker beliefs about influenza vaccine and reasons for non-vaccination--a cross-sectional survey. J Clin Nurs. 2005 Sep;14(8):922-5. doi: 10.1111/j.1365-2702.2005.01190.x. PMID 16102143
- [Background] Douville LE, Myers A, Jackson MA, Lantos JD. Health care worker knowledge, attitudes, and beliefs regarding mandatory influenza vaccination. Arch Pediatr Adolesc Med. 2010 Jan;164(1):33-7. doi: 10.1001/archpediatrics.2009.252. PMID 20048239
- [Background] van den Dool C, Bonten MJ, Hak E, Heijne JC, Wallinga J. The effects of influenza vaccination of health care workers in nursing homes: insights from a mathematical model. PLoS Med. 2008 Oct 28;5(10):e200. doi: 10.1371/journal.pmed.0050200. PMID 18959470
- [Background] Blank PR, Schwenkglenks M, Szucs TD. Vaccination coverage rates in eleven European countries during two consecutive influenza seasons. J Infect. 2009 Jun;58(6):446-58. doi: 10.1016/j.jinf.2009.04.001. Epub 2009 Apr 17. PMID 19446340
- [Background] Looijmans-van den Akker I, van Delden JJ, Verheij TJ, van der Sande MA, van Essen GA, Riphagen-Dalhuisen J, Hulscher ME, Hak E. Effects of a multi-faceted program to increase influenza vaccine uptake among health care workers in nursing homes: A cluster randomised controlled trial. Vaccine. 2010 Jul 12;28(31):5086-92. doi: 10.1016/j.vaccine.2010.05.003. Epub 2010 May 23. PMID 20580740
- [Result] Hopman CE, Riphagen-Dalhuisen J, Looijmans-van den Akker I, Frijstein G, Van der Geest-Blankert AD, Danhof-Pont MB, De Jager HJ, Bos AA, Smeets E, De Vries MJ, Gallee PM, Lenderink AF, Hak E. Determination of factors required to increase uptake of influenza vaccination among hospital-based healthcare workers. J Hosp Infect. 2011 Apr;77(4):327-31. doi: 10.1016/j.jhin.2010.10.009. Epub 2011 Feb 12. PMID 21316803
- [Derived] Meijboom MJ, Riphagen-Dalhuisen J, Hak E. The potential economic value of influenza vaccination for healthcare workers in The Netherlands. Influenza Other Respir Viruses. 2018 Jul;12(4):457-464. doi: 10.1111/irv.12558. Epub 2018 May 24. PMID 29624882
- [Derived] Riphagen-Dalhuisen J, Burgerhof JG, Frijstein G, van der Geest-Blankert AD, Danhof-Pont MB, de Jager HJ, Bos AA, Smeets EE, de Vries MJ, Gallee PM, Hak E. Hospital-based cluster randomised controlled trial to assess effects of a multi-faceted programme on influenza vaccine coverage among hospital healthcare workers and nosocomial influenza in the Netherlands, 2009 to 2011. Euro Surveill. 2013 Jun 27;18(26):20512. doi: 10.2807/1560-7917.es2013.18.26.20512. PMID 23827527
- See also: Website that was developed as part of the implementation program. — http://www.bewustgepriktvooru.nl